CLINICAL TRIAL: NCT03195140
Title: Tandem PLGS Pivotal Trial: A Randomized Clinical Trial to Assess the Efficacy of Predictive Low Glucose Suspend Versus Sensor-augmented Pump Therapy in the Management of Type 1 Diabetes
Brief Title: Diabetes Pump With Predictive Low Glucose Suspend Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G170105
Record Dates: First submitted 2017-06-14; First posted 2017-06-22 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Diabetes; Sensor Augmented Pump; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, crossover design, consisting of two 3-week periods, with the PLGS System used during one period and SAP therapy used during the other period. The crossover trial will be preceded by a run-in phase in which participants may receive training using the study devices.
  For 10 adult participants, a PLGS Pilot Period will proceed to the crossover trial to ensure safety and usability objectives are met prior to the start of the crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention Arm (Experimental): The intervention arm (use of PLGS feature) will utilize Tandem Diabetes Care's ambulatory insulin infusion pump with integrated Dexcom G5 CGM and predictive low glucose suspend function. This pump is called the "t:slim X2 with Basal-IQ Technology" and is referred to in the protocol as the Tandem PLGS pump.
  Interventions: Device: Predictive Low Glucose Suspend
- Control Arm (No Intervention): The control arm (SAP only) will utilize an identical pump in functionality as the Tandem PLGS pump except for the lack of the PLGS feature and the associated user interface. This pump is called the t:slim X2 Dexcom G5 Mobile CGM Enabled pump, and is referred to in the protocol as the Tandem SAP pump.

INTERVENTIONS:
Device: Predictive Low Glucose Suspend — Application of Predictive Low Glucose Suspend
  Arms: Intervention Arm

SUMMARY:
A 6-week crossover study will compare PLGS to SAP outcomes in adults and youth > 6 years old with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
1. Screening and Enrollment

   * Informed consent will be signed and eligibility will be assessed
   * History and physical examination
   * HbA1c measurement
   * Urine or serum pregnancy test (if applicable)
   * Evaluation of Continuous Glucose Monitoring (CGM) and pump experience
2. CGM and (Sensor Augmented Pump) SAP Training Period at Home All eligible participants will be assessed based on their CGM and pump experience to determine if the CGM Training Period, the SAP Training Period, or both are required.

   1. CGM Training Period (10-14 days): Participants currently using a CGM may skip the CGM Training Period per investigator discretion, generally requiring that CGM has been used on at least 85% of days during the prior 4 weeks.
   2. SAP Training Period (14-28 days): Participants currently using a Tandem pump concomitantly with a Dexcom CGM may skip both the CGM Training and the SAP Training periods per investigator discretion.

   i. The Tandem SAP pump will be used during the SAP Training Period and pump training will be customized based on prior pump experience
3. PLGS Pilot Phase Prior to the initiation of the crossover trial, 10 adult participants will use the Tandem PLGS pump and CGM system in a 10-day Pilot Period. Data will be evaluated for system usability and predetermined safety metrics before participants ≥12 years old can be randomized into the crossover trial.
4. Randomized Crossover Trial The crossover trial will begin after the data from the Pilot Period have been reviewed. Enrollment of participants 6 to 11 years old will be deferred until data from 100 post-randomization PLGS participant-days have been evaluated from participants 12 to 17 years old and the same predetermined safety metrics used to evaluate the Pilot Period have been satisfied.

At the Crossover Trial initiation visit, the following will be done:

* The clinician will confirm the participant's willingness to participate in the crossover trial
* The participant's HbA1c level will be measured
* Random assignment to Group A or Group B Group A: intervention period first (PLGS), control period second (SAP) Group B: control period first (SAP), intervention period second (PLGS)

During each of the two 3-week periods, a phone, email, or text contact will occur at 2 and 14 days, and a clinic visit at 7 and 21 days. HbA1c will be measured at the end of each period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis, based on investigator assessment, of T1D treated with insulin via an insulin pump or injections for at least 1 year, with no major change in the intensity of insulin therapy in the past 3 months (e.g. switching from injections to pump)
* 2. Age ≥6.0 years old
* 3. For participants <18 years old, living with one or more parents or guardians committed to participating in training and able to contact the participant in case of an emergency
* 4. For females, not currently known to be pregnant
* - If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* 5. Investigator has confidence that the participant can successfully use all study devices and is capable of adhering to the protocol

Exclusion Criteria:

* 1. Anticipated need to use acetaminophen during study participation
* 2. Participation in another pharmaceutical or device trial at the time of enrollment or plan to participate in another study during the time period of participation in this study
* 3. Employed by, or having immediate family members employed by Tandem; or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial
* 4. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk including any contraindication to the use of any of the study devices per FDA labelling
* - Individuals should not be enrolled with uncontrolled thyroid disease, renal failure (e.g., dialysis or estimated glomerular filtration (eGFR) <30), hemophilia or another major bleeding disorder, or unstable cardiovascular disease.
* - Laboratory testing and other work up needed to determine that an individual is a suitable candidate for the study should be performed as part of usual care.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University; Vance Swanson, Study Chair — Tandem Diabetes Care, Inc.; John Lum, MS, Study Director — JCHR
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - William Sansum Diabetes Center, Santa Barbara, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forlenza GP, Li Z, Buckingham BA, Pinsker JE, Cengiz E, Wadwa RP, Ekhlaspour L, Church MM, Weinzimer SA, Jost E, Marcal T, Andre C, Carria L, Swanson V, Lum JW, Kollman C, Woodall W, Beck RW. Predictive Low-Glucose Suspend Reduces Hypoglycemia in Adults, Adolescents, and Children With Type 1 Diabetes in an At-Home Randomized Crossover Study: Results of the PROLOG Trial. Diabetes Care. 2018 Oct;41(10):2155-2161. doi: 10.2337/dc18-0771. Epub 2018 Aug 8. PMID 30089663

RESULTS

PARTICIPANT FLOW:
Groups:
- PLGS First, Then SAP: Participants were randomized to use the Predictive Low-Glucose Suspend (PLGS) system first for 3 weeks, then the switch to the sensor-augmented pump (SAP) arm for 3 weeks.
- SAP First, Then PLGS: Participants were randomized to use the sensor-augmented pump (SAP) system first for 3 weeks, then the switch to the Predictive Low-Glucose Suspend (PLGS) arm for 3 weeks.
Period: Overall Study
Arm/Group | PLGS First, Then SAP | SAP First, Then PLGS
Started | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLGS First, Then SAP | SAP First, Then PLGS | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 60
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (18) | 23 (16) | 24 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 26 | 19 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 49 | 47 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 2 | 2
  White | 44 | 38 | 82
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia < 70 mg/dL
Description: Percentage of time CGM <70 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- Baseline: Measures at baseline
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 3.6 [1.9 to 5.6] | 2.6 [1.4 to 4.0] | 3.2 [1.9 to 6.1]

2. Secondary Outcome: Hypoglycemia <60 mg/dL
Description: Percentage of time CGM <60 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 1.2 [0.6 to 2.1] | 0.9 [0.4 to 1.6] | 1.2 [0.6 to 2.7]

3. Secondary Outcome: Hypoglycemia <50 mg/dL
Description: Percentage of time CGM <50 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 0.3 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.3 [0.1 to 0.7]

4. Secondary Outcome: Hypoglycemia AOC <70 mg/dL
Description: Area Over Curve (AOC) <70 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: mg*hr/dL
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
mg*hr/dL | 0.31 [0.19 to 0.55] | 0.25 [0.11 to 0.40] | 0.30 [0.17 to 0.65]

5. Secondary Outcome: Low Blood Glucose Index (LBGI)
Description: Low blood glucose index (LBGI) by CGM with higher index indicating higher risk of hypoglycemia. LBGI ≤ 1.1 is associated with minimal risk of hypoglycemia, 1.1 < LBGI ≤ 2.5 is associated with a low risk of hypoglycemia, 2.5 < LBGI ≤ 5.0 is associated with a moderate risk of hypoglycemia, and LBGI > 5.0 is associated with high risk of hypoglycemia.
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: index score
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
index score | 0.9 [0.6 to 1.3] | 0.8 [0.5 to 1.1] | 0.9 [0.6 to 1.5]

6. Secondary Outcome: Hypoglycemic Events Per Week
Description: A hypoglycemia event was defined as at least two sensor values <54 mg/dL that were ≥15 min apart with no intervening values >54 mg/dL. At least two sensor values >70 mg/dL that are ≥30 min apart with no intervening values <70 mg/dL are required to end a hypoglycemic event.
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: events/week
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
events/week | 1.1 [0.5 to 2.4] | 0.8 [0.3 to 1.9] | 1.1 [0.4 to 3.0]

7. Secondary Outcome: Time in Range 70-180 mg/dL
Description: Percentage of time CGM in range 70 to 180 mg/dL
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 64 (15) | 65 (15) | 63 (15)

8. Secondary Outcome: Hyperglycemia >250 mg/dL
Description: Percentage of time CGM >250 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 7 [3 to 15] | 8 [3 to 13] | 8 [3 to 16]

9. Secondary Outcome: Hyperglycemia >180 mg/dL
Description: Percentage of time CGM >180 mg/dL
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
percentage of time | 32 (17) | 32 (15) | 33 (16)

10. Secondary Outcome: Area Under Curve >180 mg/dL
Description: Hyperglycemia Area Under Curve of CGM >180 mg/dL
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: mg*hr/dL
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
mg*hr/dL | 14.7 [7.5 to 24.7] | 15.8 [8.3 to 24.1] | 16.9 [7.4 to 25.8]

11. Secondary Outcome: High Blood Glucose Index (HBGI)
Description: High Blood Glucose Index (HBGI) is a measure of Hyperglycemic Risk based on frequency and severity of hyperglycemic events. HBGI < 4.5 is associated with lower risk of hyperglycemia, 4.5 < HBGI < 9 is associated with a moderate risk of hyperglycemia and HBGI > 9 is associated with high risk of hyperglycemia
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: index score
Arm/Group | Baseline | Intervention Arm | Control Arm
Number analyzed (Participants) | 102 | 102 | 102
index score | 6.7 [3.9 to 9.9] | 6.9 [4.4 to 9.6] | 7.4 [4.2 to 10.1]

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Intervention Arm: The intervention arm (use of PLGS feature).
- Control Arm: The control arm (SAP only).
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103 | 2/103
Other Adverse Events (participants affected / at risk) | 58/103 | 59/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=103) | Control Arm (N=103)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=103) | Control Arm (N=103)
Ketosis (Endocrine disorders) | 58 (99) | 59 (91) — At least one day with ketones > 1.0 mmol/L

LIMITATIONS AND CAVEATS:
1 participant did not have baseline data available, so outcome measures report on 102 of the 103 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03195140/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03195140/SAP_001.pdf